CLINICAL TRIAL: NCT01994850
Title: A Phase I/II Study Of Brentuximab Vedotin In Combination With Multi-Agent Chemotherapy As Front-Line Treatment In Patients With CD30 Positive Primary Mediastinal Large B-Cell, Diffuse Large B-Cell, And Grey Zone Lymphomas
Brief Title: Brentuximab Vedotin and Chemotherapy in CD30+ PMBL, Diffuse Large B-Cell, and Grey Zone Lymphoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17413
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: CD30 Positive Primary Mediastinal Large B-cell Lymphoma; CD30-Positive Diffuse Large B-Cell Lymphoma; CD30-Positive Gray Zone Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I/II (Experimental): Total of six 21-day cycles of brentuximab vedotin in combination with rituximab, cyclophosphamide, doxorubicin and prednisone (R-CHP). Cycle 1 rituximab dose divided between Days 1 and 2 to prevent severe infusion reactions in rituximab naïve patients; brentuximab vedotin and cytotoxic chemotherapy administered on Day 2. Cycles 2 through 6 brentuximab vedotin and R-CHP administered on Day 1. Prednisone (or steroid equivalent) administered Days 1-5 of each cycle (prior to rituximab infusion).
  Cycle 1:
  Days 1-5: Prednisone (or equivalent) 100 mg PO/IV; Day 1: Rituximab 100 mg/m2 IV; Day 2: Rituximab 275 mg/m2 IV, Cyclophosphamide 750 mg/m2 IV, Doxorubicin 50 mg/m² IV, Brentuximab vedotin 1.8 mg/kg or 1.2 mg/kg (Phase I data established a MTD of 1.8 mg/kg brentuximab vedotin)
  Cycles 2-6:
  Days 1-5: Prednisone (or equivalent) 100 mg PO/IV; Day 1: Rituximab 375 mg/m2 IV, Cyclophosphamide 750 mg/m2 IV, Doxorubicin 50 mg/m² IV, Brentuximab vedotin 1.8 mg/kg
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — Trade name: Adcetris

SUMMARY:
This is a Phase I/II multicenter single arm non-randomized open label study of the investigational drug, brentuximab vedotin, given in combination with routine chemotherapy (rituximab, cyclophosphamide, doxorubicin and prednisone) every 3 weeks for a total of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Histologically confirmed CD30-positive, CD20-positive untreated primary mediastinal B-cell lymphoma (any Ann Arbor stage), diffuse large B-cell lymphoma (Ann Arbor stage III or IV), or grey zone lymphoma (any Ann Arbor stage). Patients with heterogeneous, weak or equivocal CD30 staining will also be included (no specific cut off percentage for CD30 stain is required).
* Measurable disease, defined by the Revised Response Criteria for Malignant Lymphoma
* Absolute neutrophil count ≥1,000/mmᶟ and platelet count ≥75,000/µL(unless documented bone marrow involvement with lymphoma).
* Normal left ventricular ejection fraction of ≥50% estimated by MUGA scan or echocardiogram.
* Estimated creatinine clearance (using Cockcroft-Gault equation) must be >50 mL/min.
* Serum bilirubin ≤1.5 x upper limit of normal (ULN). Bilirubin ≤ 3 x ULN is permitted in individuals with documented liver involvement by lymphoma or if due to known Gilbert syndrome.
* Aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase ≤ 3 x ULN.
* Performance status of ECOG 0-2; patients with ECOG of 3 may be allowed to enroll after discussion with the Regulatory-Sponsor/Principal Investigator and medical monitor, and if the performance status is believed to be secondary to lymphoma related symptoms and performance status is expected to improve once chemotherapy commences.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent. In patients who are not able to consent to the trial due to medical circumstances, the next of kin or power
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (b-hcG) pregnancy test result within 7 days prior to the first dose of brentuximab vedotin and must agree to use an effective contraception method during the study and for 30 days following the last dose of study drug; females of non-childbearing potential are those who are post-menopausal for more than 1 year or who have had bilateral tubal ligation or hysterectomy.
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of study drug.
* Must be able to comply with the study and follow-up requirements.

Exclusion Criteria:

* Previous use of investigational agents, chemotherapy or immunotherapy for lymphoma any time prior to enrollment (i.e. must have untreated disease). Prior allogeneic or autologous transplants are also not allowed.
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol. Consolidative radiation therapy (RT) after completion of planned course and/or concurrent intrathecal chemotherapy for CNS disease prophylaxis is permissible.
* Treatment with systemic steroids for > 4 weeks prior to Cycle 1 Day 1 of study therapy. Prior radiation therapy, with the exception of an abbreviated course (not more than 3 days) if used for SVC syndrome.
* History of serious organ dysfunction or disease involving the heart (left ventricular ejection fraction < 50%; unstable angina, acute myocardial infarction within 6 months prior to randomization, congestive heart failure NYHA III-IV, and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.), the kidney (creatinine clearance <50 mL/min), the liver (chronic hepatitis B as defined below or elevated AST, ALT or alkaline phosphatase > 3 ULN; serum bilirubin > 1.5 x ULN; bilirubin up to 3 x ULN is permitted in individuals with documented liver involvement by lymphoma or if due to known Gilbert syndrome) ot other organ system that may place the patient at undue risk to undergo treatment.
* Uncontrolled systemic fungal, bacterial, viral, or serious infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment). May be enrolled if controlled on treatment.
* Significant concurrent disease, illness or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up, or interpretation of study results.
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involved with lymphoma or stable chronic liver disease per investigator's assessment).
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
* Other malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy, with the following exceptions: Treated non-melanoma skin cancer, any in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease -free duration, are eligible for this study if definitive treatment for the condition has been completed.Organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated, or radical prostatectomy or definitive prostate irradiation has been performed.
* Positive test for the Human Immunodeficiency Virus (HIV) unless undetectable viral load within 3 months of enrollment (HIV RNA less than 48 copies/mL) and on HAART therapy.
* Positive serology for hepatitis B (HB) defined as a positive test for hepatitis B surface antigen or hepatitis B core antibody.
* Active involvement of the central nervous system (CNS) by lymphoma. Work-up for CNS involvement at diagnosis will be directed as per the treating physician and will depend on specific clinical circumstances (no brain imaging or lumbar puncture is required by this protocol).
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Svoboda, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Derived] Svoboda J, Bair SM, Landsburg DJ, Dwivedy Nasta S, Nagle SJ, Barta SK, Khan N, Filicko-O'Hara J, Gaballa S, Strelec L, Chong E, Mitnick S, Waite TS, King C, Ballard H, Youngman M, Gerson J, Plastaras JP, Maity A, Bogusz AM, Hung SS, Nakamura H, Nejati R, Steidl C, Lim M, Ruella M, Schuster SJ. Brentuximab vedotin in combination with rituximab, cyclophosphamide, doxorubicin, and prednisone as frontline treatment for patients with CD30-positive B-cell lymphomas. Haematologica. 2021 Jun 1;106(6):1705-1713. doi: 10.3324/haematol.2019.238675. PMID 32414850
- See also: Abstract: Revised response criteria for malignant lymphoma. — https://www.ncbi.nlm.nih.gov/pubmed/17242396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I/II
Started | 32
Completed | 30
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phase I/II
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 32
Lymphoma subtype [Count of Participants; unit: Participants]
  Primary Mediastinal Large B-cell Lymphoma | 23
  Diffuse Large B-Cell Lymphoma | 6
  Gray Zone Lymphoma | 2
  Not included (Subject withdrew) | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose-limiting Toxicities
Description: Dose-limiting toxicity (DLT) is any grade 3 or 4 new non-hematologic toxicity occurring during Cycle 1 requiring a dose delay of >14 days from the planned Day 1 of Cycle 2 (21 days from Day 1 of Cycle 1). The initial planned dose of brentuximab vedotin for the Phase I cohort of 6 patients is 1.8 mg/kg. This cohort will be evaluated for DLT in the first cycle of treatment. Dose de-escalation to 1.2 mg/kg will occur if ≥ 2 of 6 patients at the 1.8 mg/kg dose level experience a DLT.
Time Frame: 21 days (Cycle 1)
Population: A total of 6 subjects were evaluated for dose limiting toxicities during Phase I. Since no DLTs were observed, the Phase I subjects were included in the efficacy analysis as they received the same dose of brentuximab vedotin 1.8 mg/kg as the Phase II subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I/II
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) is defined as the proportion of patients with CR or PR according to the International Working Group Response Criteria for non-Hodgkin Lymphoma at the conclusion of systemic therapy.
Time Frame: Three to five weeks after the completion of Cycle 6 (approximately 5 months after start if treatment)
Population: 32 patients were enrolled: 1 patient withdrew, 1 was removed for protocol non-compliance, 1 was removed due to regimen violation; a total of 29 were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I/II
Number analyzed (Participants) | 29
Participants
  Complete response | 25
  Partial resonse | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the initiation of the first study treatment (Cycle 1/Day 1) to 30 days following the last administration of study treatment, which is approximately 5 months.
Arm/Group | Phase I/II
All-Cause Mortality (participants affected / at risk) | 2/31
Serious Adverse Events (participants affected / at risk) | 12/31
Other Adverse Events (participants affected / at risk) | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II (N=31)
Fever (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
MRSA bacteremia (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I/II (N=31)
Anemia (Blood and lymphatic system disorders) | 21
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Other, left ear fullness (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
other (Eye disorders) | 3 — light sensitivity, allergies, redness
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6
Gingival pain (Gastrointestinal disorders) | 2
Other (Gastrointestinal disorders) | 2 — dental plaque, tooth sensitivity
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 21
Oral dysesthesia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 9
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 3
Edema face (General disorders) | 2
Edema limbs (Gastrointestinal disorders) | 2
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 20
Fever (General disorders) | 7
Infusion related reaction (General disorders) | 4
Infusion site extravasation (General disorders) | 1
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 5
Allergic reaction (Immune system disorders) | 2
Bronchial infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 6
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 26
Neutrophil count decreased (Investigations) | 18
Platelet count decreased (Investigations) | 7
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 24
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Thrush (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 9
Dysgeusia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 11
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 19
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Hematuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Other skin irritation (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Other psoriasis (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Phlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT01994850/Prot_SAP_000.pdf